CLINICAL TRIAL: NCT00754819
Title: Colchicine Compared With Placebo to Reduce Hs-CRP in Patients With Acute Coronary Syndromes- Targeting Inflammation in Atherosclerosis Trial
Brief Title: Targeting Inflammation in Acute Coronary Syndrome Using Colchicine
Acronym: COOL
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Responsible Party: Dr John Eikelboom, McMaster University/ Hamilton Health Sciences
Organization: McMaster University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: COL0001
Record Dates: First submitted 2008-09-16; First posted 2008-09-18 (Estimated); Last update posted 2009-10-08 (Estimated); Status verified 2009-10

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Colchicine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Colchicine 1mg daily oral
  Interventions: Drug: Colchicine
- 2 (Placebo Comparator): Placebo 1 capsule daily oral
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Colchicine — 1mg once daily
  Arms: 1
Drug: Placebo — 1 capsule daily
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the effect of colchicine on high sensitivity C-reactive protein (hs-CRP), a blood marker to measure inflammation, in patients with acute coronary syndromes.

ELIGIBILITY:
Inclusion Criteria:

* All patients with a diagnosis of acute coronary syndrome who are > 18 years old and who do not have any contraindication to colchicine.

Exclusion Criteria:

* Contraindication to colchicine including any of the following:

  * hypersensitivity to colchicine
  * severe renal, hepatic or gastrointestinal disorder
  * blood dyscrasias (myelodysplasia cytopenias etc)
* Concurrent use of moderate-strong CYP3A4 inhibitors (a complete list is appended in the full protocol)
* Known severe liver disease and/or elevated transaminases > 1.5x the upper limit of normal
* Estimated GFR < 50 ml/min
* Pregnant or lactating women or women not protected by a reliable contraception method
* Current treatment with colchicine at enrollment
* Active infection or systemic inflammation eg active rheumatoid arthritis

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2008-04; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
To determine the effect of low dose colchicine on hs-CRP. | 30 days

SECONDARY OUTCOMES:
To determine the effect of colchicine on (a)platelet function and (b)short-term risk (30 days) of cardiovascular events | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: John Eikelboom, FRACP FRCPA, Study Director — McMaster University
Locations (1):
- Hamilton General Hospital, Hamilton, Ontario, Canada